CLINICAL TRIAL: NCT05644041
Title: Phase II Trial of Intravesical Gemcitabine + Docetaxel in Patients With Nonmuscle Invasive Bladder Cancer With or Without Prior Bacillus Calmette-Guérin Therapy
Brief Title: Intravesical Gem/Doce in Patients With NMIBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000198
Record Dates: First submitted 2022-11-22; First posted 2022-12-09 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Urinary Bladder Cancer
Keywords: Bacillus Calmette-Guérin (BCG); Nonmuscle invasive bladder cancer (NMIBC); Intravesical immunotherapy; Post-transurethral resection
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine induction (Experimental): Patients will receive Gemcitabine + Docetaxel once weekly for 6 weeks.
  Interventions: Drug: gemcitabine + docetaxel

INTERVENTIONS:
Drug: gemcitabine + docetaxel — The study drugs, Gemcitabine and Docetaxel, will be administered intravesically at 1000 mg and 40 mg, respectively.

SUMMARY:
Intravesical immunotherapy or chemotherapy for non-muscle invasive bladder cancer (NMIBC) is a well-established treatment for preventing or delaying tumor recurrence after tumor resection. For high-risk non-muscle invasive bladder cancer, immunotherapy in the form of intravesical Bacillus Calmette-Guérin (BCG) can be effective as first-line; nevertheless, the response rate to BCG is suboptimal with many patients failing treatment. Following BCG-failure, however, very few effective therapeutic options exist besides life-changing cystectomy. Recent shortages of BCG have pushed the use of alternative intravesical therapies for non-muscle invasive bladder cancer. At the University of Arizona Cancer Center, the use of intravesical Gemcitabine + Docetaxel (Gem/Doce) is considered as standard treatment for patients with non-invasive bladder cancer who are unable to get BCG or are BCG-resistant. The role of Gemcitabine as first-line treatment for NMIBC is poorly understood. The purpose of this study is to gain a better understanding of the use of Gemcitabine + Docetaxel intravesical chemotherapy for non-muscle invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to consent in English or Spanish; provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female ages ≥18 years.
4. Patients with intermediate or high-risk non-muscle-invasive UC of the bladder and no previous BCG treatment.

   1. Histologically confirmed intermediate or high-risk non-muscle invasive urothelial carcinoma of the bladder (Ta, T1, or Tis stage) on Transurethral Resection of Bladder Tumor (TURBT) must be obtained within 180 days of registration. OR Patients with a high-grade recurrence after 24 months since last dose of BCG.

6. Eastern Cooperative Oncology Group (ECOG) performance status Grade 0-2. 7. Post-transurethral bladder tumor resection. 8. Evidence of post-menopausal status or negative urinary pregnancy test of female pre-menopausal patients is required. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

Exclusion Criteria:

1. Known hypersensitivity reaction to gemcitabine and/or docetaxel.
2. Clinical T2 or higher stage UC of the bladder.
3. Histopathology demonstrating any small cell component, pure adenocarcinoma, pure squamous cell carcinoma, or pure CIS of the bladder.
4. Active malignancies other than the disease being treated under study.
5. Subjects with concurrent upper urinary tract (i.e. ureter, renal pelvis) urothelial carcinoma of any stage.
6. Pregnant or breast-feeding women.
7. Has an underlying substance abuse or psychiatric disorder such that, in the opinion of the investigator, the patient would be unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) for treatment with intravesical gemcitabine for patients with intermediate and high-risk NMIBC | Complete response rate will be measured at the 3-month visit
  The primary outcome measure will be CR rate, defined as the percentage of patients with CR at the 3-month visit. An event will be defined as the earliest date of recurrence as determined using the date of cystoscopy, biopsy, or cytology, whichever occurs first.

SECONDARY OUTCOMES:
Durability of response in patients who achieve CR | Duration of CR will be measured as change from the 3-month visit up to 12 months after treatment initiation
  To assess durable CR in patients who achieved CR at the 3-month visit, defined as the percentage of patients with no detectable disease 6, 9, and 12 months after treatment initiation. Duration of CR will be defined as the time from the date of evidence of CR at the 3-month visit to the earliest date of recurrence.
Tolerability and safety of the treatment | Toxicity assessment will be evaluated at the 3-month visit
  To assess adverse events using the Medical Dictionary for Regulatory Activities (MedDRA) version 21.0 and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Adverse events will be monitored during the course of treatment, and a toxicity assessment will be done after completion of treatment that will descriptively summarize any treatment-related adverse events that occur on or after the date of the first instillation of gemcitabine.
Proportion of patients who accept maintenance therapy | The assessment will be done at the 3-month visit
  To assess the number of patients who are agreeable to monthly maintenance therapy for 10 months as per patient and physician discretion.
Rate and reasons for cystectomy (if any) | Through study completion, an average of 1 year
  To assess rate of salvage cystectomy and reasons for cystectomy at the time of tumor recurrence (if any) after treatment with gemcitabine.

OTHER OUTCOMES:
Specimen collection as part of standard of care for future exploratory research | Specimens will be collected from the first TURBT (occuring between 1-3 weeks prior to treatment)
  Tissue will be collected for future exploratory analyses. Collected tissue will be stored at the University of Arizona Cancer Center Tissue Acquisition and Cellular/Molecular Analysis Shared Resource (TACMASR) for use in future studies but will not be directly assessed for the purposes of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Chipollini, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No